CLINICAL TRIAL: NCT01720121
Title: Digital Videos Disc and Printed Guidelines and Improve the Knowledge of Patients Undergoing Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: UP 4250.08
Record Dates: First submitted 2012-10-03; First posted 2012-11-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): The control group received the guidelines orientation provide by nursing team
- Guidelines printed group (Experimental): The patient received the informative material in details about the cardiac catheterization provide by the researchers
  Interventions: Other: Printed, digital video disc
- Guidelines digital video disc group (Experimental): Guidelines digital video disc group: The patient received the informative provide by digital video disc in details about the cardiac catheterization
  Interventions: Other: Printed, digital video disc

INTERVENTIONS:
Other: Printed, digital video disc — The three groups of patient received: 1)informative material in details about the cardiac catheterization provide by the researchers; 2)informative provide by a digital video disc; 3)the control group received the conventional informative provide by the nursing team.
  Arms: Guidelines digital video disc group; Guidelines printed group

SUMMARY:
This study is randomized clinical trial to verify the effect of nursing guidelines for patients undergoing left cardiac catheterization on an outpatient basis. Comparing three approaches to direct guidelines about the procedure:

* printed,
* digital video disc (DVD)
* conventional guidelines provide by nursing team

DETAILED DESCRIPTION:
This study is randomized clinical trial to verify the effect of nursing guidelines for patients undergoing left cardiac catheterization on an outpatient basis. Comparing three approaches to direct guidelines about the procedure:

* guidelines printed, (GOI) with informative material
* guidelines through a digital video disc (GDVD) six minutes
* conventional guidelines provide by nursing team

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing the procedure were included, with age equal or superior to 18 years

Exclusion Criteria:

* patients who had already undergone previous procedures similar severe comorbidities, illiterate and who came to the facility to urgently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
improvement of knowledge about the procedure after orientation | four months

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo da Silva, Professor, Principal Investigator — Federal University of Rio Grande do Sul